CLINICAL TRIAL: NCT06675942
Title: Evaluating the Short-term Efficacy of Two Oscillation Techniques in Hypersecretive Mechanically Ventilated Patients: a Randomized Crossover Trial
Brief Title: Evaluating the Short-term Efficacy of Two Oscillation Techniques in Hypersecretive Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12300126
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hypersecretive Mechanically Ventilated Patients
Keywords: Mechanical ventilation, Oscillation and Lung Expansion, High-frequency chest wall oscillation, Electrical impedance tomography
MeSH Terms: interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oscillation and Lung Expansion (Experimental)
  Interventions: Device: Oscillation and Lung Expansion; Device: High-frequency chest wall oscillation
- High-frequency chest wall oscillation (Experimental)
  Interventions: Device: Oscillation and Lung Expansion; Device: High-frequency chest wall oscillation

INTERVENTIONS:
Device: Oscillation and Lung Expansion — The OLE device (MetaNeb system) is a newer, noninvasive physiotherapy tool that combines mechanical and pharmacological interventions (aerosols) to help mobilize endobronchial secretions.
Device: High-frequency chest wall oscillation — High-frequency chest wall oscillation (HFCWO) is an airway clearance technique that uses external forces applied to the chest via an inflatable vest connected to a device that generates vibrations at varying frequencies and pressures.

SUMMARY:
Although mechanical ventilation (MV) is life-saving, it is associated with several complications. The establishment of an artificial airway impairs the cough reflex and mucociliary function, leading to the accumulation of secretions in the tracheobronchial tree. This increases the risk of pneumonia and lung atelectasis. Usual care for mechanically ventilated patients includes airway suctioning via the tracheostomy tube, which clears only a limited portion of the airway and is ineffective at removing peripheral airway secretions.

To address this, airway clearance guidelines recommend various airway clearance techniques (ACTs) for mechanically ventilated patients to enhance mucus removal. However, the lack of standardized, effective evaluation criteria makes selecting the optimal ACT a challenge.

DETAILED DESCRIPTION:
The aim of this randomized cross-over study was to compare the effectiveness of oscillation and lung expansion (OLE) versus high-frequency chest wall oscillation (HFCWO) on lung aeration and ventilation distribution, as assessed by EIT, in medically complex, hypersecretive patients with tracheostomy tubes requiring long-term mechanical ventilation (MV).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were patients aged ≥18 years with airway hypersecretion, admitted to the ICU,
* Requiring more than 48 hours of MV.

Exclusion Criteria:

* Malignant arrhythmia
* Acute myocardial ischemia
* Pneumothorax, pulmonary bulla, barotrauma, or other lung diseases,
* Hemorrhagic disease or coagulation abnormalities with bleeding tendencies
* Skin trauma on the chest
* Pulmonary embolism
* Presence of a permanent or temporary pacemaker
* Untreated spinal and rib fractures
* Any condition deemed inappropriate for study inclusion by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
End-expiratory lung impedance (EELI) | at the end of treatment (T1) and at 1 hour (T2), 2 hours (T3), 4 hours (T4)

SECONDARY OUTCOMES:
Tidal impedance variation (TV) | at the end of treatment (T1) and at 1 hour (T2), 2 hours (T3), 4 hours (T4)
sputum volume | at the end of treatment (T1) and at 1 hour (T2), 2 hours (T3), 4 hours (T4)
Respiratory rate | at the end of treatment (T1) and at 1 hour (T2), 2 hours (T3), 4 hours (T4)
center of ventilation (COV) | at the end of treatment (T1) and at 1 hour (T2), 2 hours (T3), 4 hours (T4)

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ge, Principal Investigator — Beijing Rehabilitation Hospital of Capital Medical University
Locations (1):
- Beijing Rehabilitation Hospital, Beijing, China